CLINICAL TRIAL: NCT00641849
Title: Physical Activity and Dietary Behaviors of Adults 18 to 80 Years of Age
Acronym: Compliance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by PI r/t lack of funding and retirement of study personel.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1103057
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Physical Activity
Keywords: BMI; Physical Activity; Food; Nutrition; Dietary behaviors; Diet; Adult; Adults; Fat; Fats; Self monitoring; Automated feedback
MeSH Terms: conditions — Motor Activity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Minimum Intervention Group A will fill out data forms at zero (0), two (2), four (4), and six (6) months.
  Interventions: Behavioral: Group A
- Group B (Active Comparator): Maximum Intervention Group B will fill out data forms at zero (0), one (1), two (2), three (3), four (4), five (5), and six (6) months.
  Interventions: Behavioral: Group B

INTERVENTIONS:
Behavioral: Group A — Minimum Intervention Group A will fill out data forms at zero (0), two (2), four (4), and six (6) months.
  Other Names: Minimal intervention
  Arms: Group A
Behavioral: Group B — Maximum Intervention Group B will fill out data forms at zero (0), one (1), two (2), three (3), four (4), five (5), and six (6) months.
  Other Names: Maximum intervention
  Arms: Group B

SUMMARY:
This research will focus on the effect of a 6-month behavioral intervention delivered via the World Wide Web that is aimed at increasing physical activity levels and decreasing dietary fat intake in a general population of adults. The study will be randomized and blinded. We are also planning to study subjects' compliance and retention rates when enrolled in a completely on-line study.

DETAILED DESCRIPTION:
The research is designed as a prospective multi-site, randomized, blinded trial.

Participants will fill out an initial questionnaire 72 hours (time 0) after completing the inclusion/exclusion questionnaire and consent documents. An email will be sent sixty (60) hours after participants who agreed to the online consent and HIPAA articles. Subjects who have consented to participate in the trial will not be considered as enrolled until after they have completed their time 0 data forms and completed the education module.

The subjects will be randomly assigned to either the minimum or maximum treatment group. Both groups will be sent an email reminder 7 days prior to their "follow-up" date. They will then be sent an email reminder 24 hours prior to their "follow-up" date. Subjects will receive an email reminder every 48 hours until 336 hours (14 days) post visit date. Reminder emails will also state that those subjects not completing their "follow-up" visit within the visit window will be withdrawn from the study. Subjects will be not be blinded as to how frequently they will be required to make "follow-up" visits to the site.

Group A: Minimum Intervention Group A will fill out data forms at zero (0), two (2), four (4), and six (6) months.

Group B: Maximum Intervention Group B will fill out data forms at zero (0), one (1), two (2), three (3), four (4), five (5), and six (6) months.

A short online education module will be given after the initial surveys (time 0) have been completed by the study subject. They will receive their initial "feedback" letter after completing the education module. It will also tell them the date of their "follow-up" visit, and that they will be periodically prompted to return to the site and complete a questionnaire.

Both groups will receive a "feedback" letter upon completion of each online "follow-up" visit. This letter will give them "feedback" based off of how they answered their data forms. All "feedback" given will be based off of established recommended physical activity and the USDA food pyramid guidelines. The BMI will be calculated; BMI = weight (kg)/height2 (m2).

Subjects in both groups who have not completed their "follow-up" visits after 336 hours (14 days) post visit date will be sent an email notifying them that they have been dropped from the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years to 80 years
* Participants must be willing to complete initial questionnaire 72 hours after completing inclusion criteria screening and review of informed consent
* Participants must be willing to review educational module
* Participants must be willing to fill out seven (7) questionnaires per protocol.

Exclusion Criteria:

-Individuals who do not have access to the Internet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the level of compliance and retention between the two groups. | Six months

SECONDARY OUTCOMES:
Mean physical activity levels of trial completers relative to their mean baseline PA levels. | Six months
Mean fat intake score of trial completers relative to their mean baseline fat intake. | Six months
Mean body mass index (BM) of trial completers relative to their mean baseline BMI. | Six Months
Comparison of mean physical activity level, fat intake scores, and BMI of trial completers in each treatment arm at 6 months (outcome means adjusted for baseline values). | Six months
Changes in PA levels, fat intake scores and BMI over time for subjects in each treatment arm. | Six months
Intent-to treat analysis will be conducted at outcome for physical activity, fat intake scores and BMI by carrying the last entered values forward to represent the values at outcome. Intent to treat analysis may be precluded by a high dropout rate. | Six months
Subject reported satisfaction with participation in an on-line study | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Cooper, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Northern Arizona University, Flagstaff, Arizona
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauman AE. Updating the evidence that physical activity is good for health: an epidemiological review 2000-2003. J Sci Med Sport. 2004 Apr;7(1 Suppl):6-19. doi: 10.1016/s1440-2440(04)80273-1. PMID 15214597
- [Background] Pfohl M, Schatz H. Strategies for the prevention of type 2 diabetes. Exp Clin Endocrinol Diabetes. 2001;109 Suppl 2:S240-9. doi: 10.1055/s-2001-18585. PMID 11460574
- [Background] Wannamethee SG, Shaper AG. Physical activity in the prevention of cardiovascular disease: an epidemiological perspective. Sports Med. 2001 Feb;31(2):101-14. doi: 10.2165/00007256-200131020-00003. PMID 11227978
- [Background] Gorelick PB, Sacco RL, Smith DB, Alberts M, Mustone-Alexander L, Rader D, Ross JL, Raps E, Ozer MN, Brass LM, Malone ME, Goldberg S, Booss J, Hanley DF, Toole JF, Greengold NL, Rhew DC. Prevention of a first stroke: a review of guidelines and a multidisciplinary consensus statement from the National Stroke Association. JAMA. 1999 Mar 24-31;281(12):1112-20. doi: 10.1001/jama.281.12.1112. PMID 10188663
- [Background] Kuller LH. Dietary fat and chronic diseases: epidemiologic overview. J Am Diet Assoc. 1997 Jul;97(7 Suppl):S9-15. doi: 10.1016/s0002-8223(97)00724-4. PMID 9216562
- [Background] U.S. Dept of Health and Human Services: Physical Actvity and Health: A report of the Sugeon General. Atlanta GA: Centers for Disease Control and Prevention, National Center for Chronic Deases Prevention and Health Promotion 1996.
- [Background] Physical activity and cardiovascular health. NIH Consens Statement. 1995 Dec 18-20;13(3):1-33. PMID 9160011
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] National Center for Health Statistics. National Health Interview Survey, 2005: Hyattsville MD: National Center for Health Statistics, 2007.
- [Background] U.S. Department of Health and Human Services. Healthy People 2010: National health promotion and disease prevention objectives. Washington DC: U.S Department of Health and Human Services 2000.
- [Background] Ammerman AS, Lindquist CH, Lohr KN, Hersey J. The efficacy of behavioral interventions to modify dietary fat and fruit and vegetable intake: a review of the evidence. Prev Med. 2002 Jul;35(1):25-41. doi: 10.1006/pmed.2002.1028. PMID 12079438
- [Background] Kahn EB, Ramsey LT, Brownson RC, Heath GW, Howze EH, Powell KE, Stone EJ, Rajab MW, Corso P. The effectiveness of interventions to increase physical activity. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):73-107. doi: 10.1016/s0749-3797(02)00434-8. PMID 11985936
- [Background] Sherwood NE, Jeffery RW. The behavioral determinants of exercise: implications for physical activity interventions. Annu Rev Nutr. 2000;20:21-44. doi: 10.1146/annurev.nutr.20.1.21. PMID 10940325
- [Background] Gillman MW, Pinto BM, Tennstedt S, Glanz K, Marcus B, Friedman RH. Relationships of physical activity with dietary behaviors among adults. Prev Med. 2001 Mar;32(3):295-301. doi: 10.1006/pmed.2000.0812. PMID 11277687
- [Background] Eaton CB, McPhillips JB, Gans KM, Garber CE, Assaf AR, Lasater TM, Carleton RA. Cross-sectional relationship between diet and physical activity in two southeastern New England communities. Am J Prev Med. 1995 Jul-Aug;11(4):238-44. PMID 7495600
- [Background] AbuSabha R, Achterberg C. Review of self-efficacy and locus of control for nutrition- and health-related behavior. J Am Diet Assoc. 1997 Oct;97(10):1122-32. doi: 10.1016/S0002-8223(97)00273-3. PMID 9336559
- [Background] Marcus BH, Lewis BA, Williams DM, Dunsiger S, Jakicic JM, Whiteley JA, Albrecht AE, Napolitano MA, Bock BC, Tate DF, Sciamanna CN, Parisi AF. A comparison of Internet and print-based physical activity interventions. Arch Intern Med. 2007 May 14;167(9):944-9. doi: 10.1001/archinte.167.9.944. PMID 17502536
- [Background] Tate DF, Jackvony EH, Wing RR. A randomized trial comparing human e-mail counseling, computer-automated tailored counseling, and no counseling in an Internet weight loss program. Arch Intern Med. 2006 Aug 14-28;166(15):1620-5. doi: 10.1001/archinte.166.15.1620. PMID 16908795
- [Background] Armitage CJ, Conner M. Efficacy of a minimal intervention to reduce fat intake. Soc Sci Med. 2001 May;52(10):1517-24. doi: 10.1016/s0277-9536(00)00265-3. PMID 11314848
- [Background] Marcus BH, Bock BC, Pinto BM, Forsyth LH, Roberts MB, Traficante RM. Efficacy of an individualized, motivationally-tailored physical activity intervention. Ann Behav Med. 1998 Summer;20(3):174-80. doi: 10.1007/BF02884958. PMID 9989324
- [Background] Marcus BH, Emmons KM, Simkin-Silverman LR, Linnan LA, Taylor ER, Bock BC, Roberts MB, Rossi JS, Abrams DB. Evaluation of motivationally tailored vs. standard self-help physical activity interventions at the workplace. Am J Health Promot. 1998 Mar-Apr;12(4):246-53. doi: 10.4278/0890-1171-12.4.246. PMID 10178617
- [Background] Brug J, Steenhuis I, van Assema P, de Vries H. The impact of a computer-tailored nutrition intervention. Prev Med. 1996 May-Jun;25(3):236-42. doi: 10.1006/pmed.1996.0052. PMID 8781000
- [Background] Cook RF, Billings DW, Hersch RK, Back AS, Hendrickson A. A field test of a web-based workplace health promotion program to improve dietary practices, reduce stress, and increase physical activity: randomized controlled trial. J Med Internet Res. 2007 Jun 19;9(2):e17. doi: 10.2196/jmir.9.2.e17. PMID 17581811
- [Background] McKay HG, King D, Eakin EG, Seeley JR, Glasgow RE. The diabetes network internet-based physical activity intervention: a randomized pilot study. Diabetes Care. 2001 Aug;24(8):1328-34. doi: 10.2337/diacare.24.8.1328. PMID 11473065
- [Background] Marcus BH, Nigg CR, Riebe D, Forsyth LH. Interactive communication strategies: implications for population-based physical-activity promotion. Am J Prev Med. 2000 Aug;19(2):121-6. doi: 10.1016/s0749-3797(00)00186-0. PMID 10913903
- [Background] Kroeze W, Werkman A, Brug J. A systematic review of randomized trials on the effectiveness of computer-tailored education on physical activity and dietary behaviors. Ann Behav Med. 2006 Jun;31(3):205-23. doi: 10.1207/s15324796abm3103_2. PMID 16700634
- [Background] Spittaels H, De Bourdeaudhuij I, Vandelanotte C. Evaluation of a website-delivered computer-tailored intervention for increasing physical activity in the general population. Prev Med. 2007 Mar;44(3):209-17. doi: 10.1016/j.ypmed.2006.11.010. Epub 2007 Jan 2. PMID 17197015
- [Background] Harvey-Berino J, Pintauro S, Buzzell P, DiGiulio M, Casey Gold B, Moldovan C, Ramirez E. Does using the Internet facilitate the maintenance of weight loss? Int J Obes Relat Metab Disord. 2002 Sep;26(9):1254-60. doi: 10.1038/sj.ijo.0802051. PMID 12187404
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Appendix B22. Dietary Quality: The Food Habits Questionnaire. In: St. Jeor ST, ed. Obesity Assessment: Tools, Methods, Interpretations. New York: Chapman & Hall, 1997, 806-812.
- [Background] Silverstein LJ, Scott BJ, Zahrt H. Dietary Quality: The Food Habits Questionnaire. In: St. Jeor ST, ed. Obesity Assessment: Tools, Methods, Interpretations. New York: Chapman & Hall; 1997: 281-291.
- See also: 7.2.4.3 Sample Size Required." Engineering Statistics Handbook, National Institute of Standards and Technology. 28 February 2008 — http://www.itl.nist.gov/div898/handbook/prc/section2/prc222.htm